CLINICAL TRIAL: NCT01419158
Title: Targeted Detection of Alpha-1 Antitrypsin Deficiency in Patients Referred for Pulmonary Function Testing
Brief Title: Prevalence of Alpha-1 Antitrypsin Deficiency in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: PFT
Status: Completed | Type: Observational
Sponsor: Alpha-1 Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PFT-001
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-09

CONDITIONS: Alpha-1 Antitrypsin Deficiency; Chronic Obstructive Pulmonary Disease
Keywords: Alpha-1 antitrypsin; Alpha-1 antitrypsin deficiency; Chronic obstructive pulmonary disease
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Alpha-1 antitrypsin deficiency (AATD) is considered a rare genetic cause of chronic obstructive pulmonary disease (COPD) and liver disease. Recent data has suggested that AATD is not as rare as originally thought and undetected AATD may account for COPD in some patients. This study was designed to evaluate the frequency of undetected AATD in a population reporting to academic pulmonary function testing facilities who meet criteria for the diagnosis of COPD. All individuals meeting GOLD criteria for COPD will be consented and offered free testing for AATD. The results will help identify the percent of those with COPD who have undetected AATD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults at least 18 years of age able to understand and consent to the procedures of this protocol.
* All races and ethnicities will be considered for this study.
* Post-bronchodilator values for pulmonary function tests on the day of enrollment with an FEV1 < 80% of predicted and FEV1/FVC < 70% (at least GOLD stage II).
* Subjects who have been tested for Alpha-1 in the past but do not know their genotype or phenotype may be included in this study.

Note: For the inclusion criteria the investigators will use the patient's GOLD status, based on percent predicted (FEV1 < 80% of predicted); however, after sending the absolute value of FEV1 to the Data Coordinating Center (DCC) the DCC will calculate the percent predicted using a standardized formula (NHANES III). For sites that do not use this predicted formula, the results obtained at the DCC may differ from those used for subject enrollment. (For example, a subject found to have an FEV1 of <80% at the study site could have an FEV1 > 80% when the DCC recalculates it). Enrollment will be based on the percent predicted at each study site. If necessary, the data from this small number of outliers will be analyzed separately.

Exclusion Criteria:

* Subjects in whom post-bronchodilator spirometry is not performed.
* Subjects whose ordering physician has specifically requested that his patients not be considered for enrollment.
* Patients who have been tested for Alpha-1 in the past and know their genotype or phenotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals reporting for pulmonary function testing who meet criteria for the diagnosis of chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 3457 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Sandhaus, M.D., Ph.D., Principal Investigator — National Jewish Health
Locations (19):
- United States (18):
  - University of California Los Angeles, Los Angeles, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Florida (Gainesville), Gainesville, Florida
  - University of Florida (Jacksonville), Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Miami VA Medical Center, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Luke's-Roosevelt Hospital Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center at Tyler, Tyler, Texas
- San Juan City Hospital, Centro Medico Metropolitano, San Juan, Puerto Rico